CLINICAL TRIAL: NCT05061277
Title: A PHASE 1, OPEN-LABEL, SINGLE SUBCUTANEOUS DOSE STUDY TO EVALUATE THE PHARMACOKINETICS, SAFETY AND TOLERABILITY OF LYOPHILIZED FORMULATION OF RECIFERCEPT IN HEALTHY CHINESE PARTICIPANTS
Brief Title: Study to Evaluate the Pharmacokinetics, Safety and Tolerability of Recifercept in Healthy Chinese Participants
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Pfizer has decided to cancel study C4181006 due to strategic considerations. This decision is not due to any specific reasons or requests from any regulatory authorities. No participants have been enrolled in this study.
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: C4181006
Record Dates: First submitted 2021-09-20; First posted 2021-09-29 (Actual); Last update posted 2023-04-18 (Actual); Status verified 2023-04

CONDITIONS: Healthy

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Recifercept (Experimental): A 300 mg single subcutaneous (SC) dose of recifercept for the treatment phase of study
  Interventions: Drug: Recifercept

INTERVENTIONS:
Drug: Recifercept — A lyophilized powder for solution for injection
  Other Names: PF-07256472

SUMMARY:
The purpose of this study is to evaluate the pharmacokinetic (PK), safety, tolerability and immunogenicity of a single subcutaneous (SC) dose of the lyophilized formulation of recifercept in healthy Chinese participants.

ELIGIBILITY:
Inclusion Criteria:

* Chinese male and female participants of nonchildbearing potential must be 21 to 55 years of age, inclusive at the time of signing the ICD.
* Chinese male and female participants who are overtly healthy as determined by medical evaluation.
* Participants who are willing and able to comply with all scheduled visits, treatment plan, laboratory tests, lifestyle considerations, and other study procedures.
* Participants must be of Chinese ethnicity (individuals currently residing in mainland China who were born in China and have both parents of Chinese descent).
* Body mass index (BMI) of 19.0 to 27.5 kg/m2; and a total body weight >50 kg and ≤ 120 kg.
* Capable of giving signed informed consent, which includes compliance with the requirements and restrictions listed in the ICD and in this protocol.

Exclusion Criteria:

* Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurological, or allergic disease (including drug allergies, but excluding untreated, asymptomatic, seasonal allergies at the time of dosing).
* Any condition possibly affecting drug absorption (eg, skin inflammation at infusion site, acne, rash, scarring, tattoos, erythema, sunburn, deep tanning, etc).
* History of human immunodeficiency virus (HIV) infection, hepatitis B, or hepatitis C; positive testing for HIV, hepatitis B surface antigen (HBsAg), hepatitis C antibody (HCVAb), or serological reaction of syphilis. Prior hepatitis B vaccination is allowed.
* Other medical or psychiatric condition including recent (within the past year) or active suicidal ideation/behavior or laboratory abnormality that may increase the risk of study participation or, in the investigator's judgment, make the participant inappropriate for the study.
* Use of prescription or nonprescription drugs and dietary and herbal supplements within 7 days or 5 half lives (whichever is longer) prior to the dose of study intervention.
* Previous administration with an investigational drug/medical device within 30 days (or as determined by the local requirement) or 5 half lives preceding the dose of study intervention used in this study (whichever is longer).
* A positive urine drug test.
* Screening supine blood pressure (BP) ≥140 mm Hg (systolic) or ≥90 mm Hg (diastolic), following at least 5 minutes of supine rest. Pulse rate > 100 beats/minute. Oral temperature (or ear temperature) > 37.5 ℃.
* Baseline 12 lead ECG that demonstrates clinically relevant abnormalities that may affect participant safety or interpretation of study results (eg, baseline corrected QT (QTc) interval >450 msec, complete LBBB, signs of an acute or indeterminate age myocardial infarction, ST T interval changes suggestive of myocardial ischemia, second or third degree AV block, or serious bradyarrhythmias or tachyarrhythmias).
* Participants with ANY of the following abnormalities in clinical laboratory tests at Screening, as assessed by the study specific laboratory and confirmed by a single repeat test, if deemed necessary:

  * aspartate aminotransferase (AST) or aspartate aminotransferase (ALT) level ≥ 1.5 × upper limit of normal (ULN);
  * Total bilirubin level ≥1.5 × ULN; participants with a history of Gilbert's syndrome may have direct bilirubin measured and would be eligible for this study provided the direct bilirubin level is≤ ULN.

Ages: 21 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2023-10-25 (Estimated); Primary Completion 2023-12-12 (Estimated); Study Completion 2024-06-16 (Estimated)

PRIMARY OUTCOMES:
Maximum Observed Concentration (Cmax) | 0, 2, 4, 6, 12, 24, 48, 72, 120, 168, 216, 264, 312, 504 hours post-dose
Time for Cmax (Tmax) | 0, 2, 4, 6, 12, 24, 48, 72, 120, 168, 216, 264, 312, 504 hours post-dose
Area Under the Serum Concentration Time Profile from Time Zero to 168 hrs (AUC0-168) | 0, 2, 4, 6, 12, 24, 48, 72, 120, 168 hours post-dose
Area Under the Serum Concentration-Time Profile From Time 0 to the Time of the Last Quantifiable Concentration (AUClast) | 0, 2, 4, 6, 12, 24, 48, 72, 120, 168, 216, 264, 312, 504 hours post-dose
Area Under the Serum Concentration Time Profile from Time 0 Extrapolated to Infinite Time (AUCinf) | 0, 2, 4, 6, 12, 24, 48, 72, 120, 168, 216, 264, 312, 504 hours post-dose
Terminal Elimination Half-Life (t½) | 0, 2, 4, 6, 12, 24, 48, 72, 120, 168, 216, 264, 312, 504 hours post-dose
Apparent Clearance (CL/F) | 0, 2, 4, 6, 12, 24, 48, 72, 120, 168, 216, 264, 312, 504 hours post-dose
Apparent Volume of Distribution (Vz/F) | 0, 2, 4, 6, 12, 24, 48, 72, 120, 168, 216, 264, 312, 504 hours post-dose

SECONDARY OUTCOMES:
Incidence of Participants With Positive Anti-Drug Antibodies (ADA) | 0, 168, 312, 504, 672 hours post-dose and maybe months 4 and/or month 7 post-dose
Incidence of Participants With Positive Neutralizing Antibodies (NAb) | Maybe 0, 168, 312, 504, 672 hours post-dose and maybe months 4 and/or month 7 post-dose
Incidence of Adverse Events (AEs) | Since inform consent form (ICD) is signed till up to about Day 29, or maybe till Month 4 or Month 7 post-dose, or when terminated/withdrawal from study
Incidence of Clinical Laboratory Test Abnormalitiests | Baseline to approximately Day 22, or up to approximately Month 4 or Month 7 post-dose, or when terminated/withwal from study
Incidence of Participants With Clinically Relevant Changes in Vital Signs | Baseline, within -3 hours pre-dose, and at 4, 24, 48, 72 hours post-dose, or up to approximately Month 4 or Month 7 post-dose, or when terminated/withdrawal from study
Incidence of Participants With Clinically Relevant Changes in 12-lead Electrocardiogram (ECG) | Baseline, within -3 hours pre-dose, and at 4, 24, 48, 72 hours post-dose, or up to approximately Month 4 or Month 7 post-dose, or when terminated/withdrawal from study
Incidence of Participants With Infusion Site Reactions | From time of signing inform concent form (ICD) to approximately Day 29, or up to approximately Month 4 or Month 7 post-dose, or when terminated/withdrawal from study

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Huashan Hospital Fudan University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C4181006